CLINICAL TRIAL: NCT05870163
Title: A Post-market Registry Study to Assess Safety and Performance of RefluxStop™ in the Treatment of Gastroesophageal Reflux Disease (GERD) in General Hospital Practice
Brief Title: Post-Market Registry for the Evaluation of RefluxStop in GERD Treatment
Status: Recruiting | Type: Observational
Sponsor: Implantica CE Reflux Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: RXI002
Record Dates: First submitted 2023-04-14; First posted 2023-05-23 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Gastroesophageal Reflux Disease (GERD)
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Fundoplication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- RefluxStop patients
  Interventions: Device: RefluxStop implantation
- Nissen fundoplication patients
  Interventions: Procedure: Nissen fundoplication

INTERVENTIONS:
Device: RefluxStop implantation — Standard surgical technique for implantation RefluxStop, as described in the Itructions for Use
  Groups: RefluxStop patients
Procedure: Nissen fundoplication — Standard of care Nissen fundoplication surgery
  Groups: Nissen fundoplication patients

SUMMARY:
This post-market registry aims to assess safety and performance of RefluxStop™ in the treatment of Gastroesophageal Reflux Disease (GERD) in standard of care procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide informed consent and to participate in the registry study,
2. Patient's age ≥ 18 years or according to local legal age of adulthood if older,
3. Documented GERD present for > 6 months,
4. Patient has a 24-hour pH monitoring proven GERD with pH and/or impedance pH measurement, off PPI therapy for at least 7 days prior to testing. (Total distal esophageal pH must be <4 for >4.5% of time during a 24-hour monitoring and/or total reflux episodes of acid >55 or weakly acid >26 for >5 seconds at 5 cm above LES)
5. Suitable to undergo general anesthesia and is a suitable laparoscopic surgery candidate as determined by the investigator.

Exclusion criteria:

1. Presence of para-esophageal hernia or sliding hernia > 3 centimeters,
2. Known presence of delayed gastric emptying, if no other cause for acid reflux could be diagnosed,
3. History of bariatric surgery wherein the stomach fundus has been extirpated,
4. Female patients who are pregnant or nursing,
5. Known sensitivity or allergies to silicone materials,
6. Intraoperative findings determined by the investigator that may result in unfavorable conduct of the registry study procedure (as outlined in the IFU);
7. Patients that are unable to comply with the registry study requirements, (for example due to major psychiatric disorder or are considered otherwise unsuitable for participation in the registry study according to the investigator's judgement).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: RefluxStop device and Nissen fundoplication are indicated for patients diagnosed with Gastroesophageal Reflux Disease (GERD) defined by abnormal pH testing.
Sampling Method: Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2023-02-20 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary safety endpoint | 6 months
  Incidence of Serious Adverse Device Effects (SADEs), Serious Adverse Events (SAEs) and Device Deficiencies (DDs)
Primary performance endpoint | 6 months
  Assessment of GERD symptoms, measured by GERD Health-Related Quality of Life (HRQL) score (questions 1-10).
  (An answer of zero means no symptoms)

SECONDARY OUTCOMES:
Secondary safety endpoint | 3 and 6 months and annually up to 5 years
  Incidence of Serious Adverse Device Effects (SADEs), Serious Adverse Events (SAEs) and Device Deficiencies (DDs) at 3 months and annually up to 5 years.
  Plus Incidence of Adverse Device Effects (ADEs) and procedure related or unknown Adverse Events (AEs) at 3 and 6 months and annually up to 5 years
Secondary performance endpoints | 3 months and annually up to 5 years
  Assessment of GERD symptoms, assessed by GERD-HRQL score (questions 1-10)
Secondary performance endpoints: RefluxStop device position | 6 months
  Location and function of the device evaluated by a simplified contrast swallow x-ray with overview pictures of device
Secondary performance endpoints: hernia assessment | 6 months
  Location of baseline hernia or any new hernia by a simplified contrast swallow x-ray picture
Secondary performance endpoints: pH monitoring | 6 months
  Reduction or normalisation from baseline of the total acid (pH<4) exposure time during 24-hour pH monitoring

OTHER OUTCOMES:
Exploratory endpoints: Patient Reported Outcomes - Quality of life questionnaire | 3 and 6 months and annually up to 5 years
  EQ-5D (Euro Quality of life-5 Dimension) questionnaire: measure of quality of life with one question for each of the five dimensions that are mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. For each dimension, the patients assess if they have no problem, slight, moderate, severe or extreme problems.
Exploratory endpoints: Patient Reported Outcomes - Work related questionnaire | 3 and 6 months and annually up to 5 years
  WPAI (work related productivity gains): 5 questions to assess how health problems effect the patient work Score 0 to 10. Zero meaning health problems have no effect on work
Exploratory endpoints: Health economic outcomes - Visit to General Practitioner | 3 and 6 months and annually up to 5 years
  Evaluation of number of visit to the General Practitioner
Exploratory endpoints: Health economic outcomes - PPI treatment use | 3 and 6 months and annually up to 5 years
  Counting of the number of patients using PPI (Proton Pump Inhibitors)
Exploratory endpoints: Health economic outcomes - Re-admission to hospital | 3 and 6 months and annually up to 5 years
  Counting of the number of re-admission to hospital due to complications
Exploratory endpoints: Health economic outcomes - Procedure costs | 3 and 6 months and annually up to 5 years
  Evaluation of the costs related to the study procedure and the length of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Yves Borbély, Dr. med., Principal Investigator — Inselspital, Universitätsspital Bern
Locations (6):
- Klinikum Friedrichshafen GmbH, Friedrichshafen, Germany
- Italy (2):
  - Ospedale IRCCS Saverio De Bellis, Bari
  - Ospedale Buon Consiglio Fatebenefratelli, Napoli
- Akershus Universitetssykehus HF, Lørenskog, Norway
- Switzerland (2):
  - Inselspital, Universitätsspital Bern, Bern
  - Hirslanden Klinik, Bern

IPD SHARING:
Plan to Share IPD: No